CLINICAL TRIAL: NCT04169984
Title: Myofunctional Therapy in Patients With Mild-moderate Sleep Apnea. Randomized Clinical Trial (MYTOSA).
Brief Title: Myofunctional Therapy in Patients With Mild-moderate Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Irene Cano-Pumarega, Principal Investigator, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYTOSA
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea of Adult; Myofunctional Therapy
MeSH Terms: interventions — Myofunctional Therapy

STUDY DESIGN:
Intervention Model Description: Two arms: active treatment group (myofunctional therapy) and placebo group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofunctional Therapy (Active Comparator): This therapy consists of the practice of isotonic, isokinetic and isometric exercises that improve mobility and coordination and increase the muscular strength of the orofacial structures that contribute to the obstructive sleep apnea etiopathogenesis.
  Interventions: Other: Myofunctional Therapy
- Placebo (Placebo Comparator): The placebo group will be instructed in simulation exercises that do not alter the function or morphology of the upper airway.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Myofunctional Therapy — Isometric, isokinetic and isotonic exercises for the upper airway muscles.
  Arms: Myofunctional Therapy
Other: Placebo — Exercises that do not alter the function or morphology of the upper airway.
  Arms: Placebo

SUMMARY:
The main objective of this study is to compare the change in the apnea-hypopnea index (AHI) in patients with mild to moderate sleep apnea without daytime sleepiness after 12 months of myofunctional therapy exercises with respect to the placebo group (the placebo group will be instructed in simulation exercises that do not alter the function or morphology of the upper airway)

DETAILED DESCRIPTION:
Background: Alternative treatment therapies to positive upper airway pressure (CPAP) for obstructive sleep apnea syndrome (OSAS) have been developed in recent years. Myofunctional orofacial therapy (MFT) is one of these alternatives and consists of exercises that improve mobility and increase muscle strength of the orofacial structures that contribute to the etiopathogenesis of OSAS. To date, any study to treat sleep apnea patients under this therapy has been conducted in Spain. Moreover, its long-term effect has not been evaluated worldwide.

Main objective: to compare the reduction in the apnea-hypopnea index (AHI) in patients with mild to moderate sleep apnea without daytime sleepiness after 12 months of myofunctional therapy exercises with respect to the placebo group (the placebo group will be instructed in simulation exercises that do not alter the function or morphology of the upper airway) Methodology: A 12-month, randomized, parallel-group, clinical trial will be conducted. Patients with an AHI ≥ 5 events per hour assessed by a respiratory polygraphy (RP) will be randomized to a MFT treatment branch or to another placebo exercises branch. A speech therapist will instruct patients to perform the exercises in both groups for three months. At the end of this period, a RP will be performed on both groups and the same treatment that they were doing will be maintained at home. One year later, a new RP will be performed and changes in AHI, oximetry parameters and snoring will be compared in both groups, as well as sleepiness, quality of life and the degree of adherence to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 80 years old.
* Patients with apnea-hypopnea index from 5 to 29 assessed by a respiratory polygraphy.
* Absence of daytime sleepiness (Epworth sleepiness scale <12).

Exclusion Criteria:

* Refractory high blood pressure (blood pressure that is not controlled with three antihypertensive drugs, including a diuretic).
* Ictus, transient ischemic attack, neuromuscular diseases, acute coronary syndrome or hospitalization for worsening heart failure, in the previous 30 days.
* Professional drivers, profession of risk or respiratory failure.
* Previous surgical intervention for the treatment of sleep apnea (those patients who have refused treatment with CPAP or mandibular advancement devices after 1 month of not using them,could be included).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in AHI after myofunctional therapy | 3 months;12 months
  To compare the apnea-hypopnea index (AHI) in patients with mild to moderate sleep apnea without daytime sleepiness after 12 months of myofunctional therapy exercises with respect to the placebo group.

SECONDARY OUTCOMES:
Change in AIH after 1 year of myofunctional treatment compared to 3 months | 3 months;12 months
  To assess whether the change in IAH is maintained comparing 12 months of active home treatment with 3 months of active treatment with a speech pathologist.
Change in snoring | 3 months;12 months
  To assess the change in snoring measured by the average intensity in decibels and the number of snoring events per hour.
Change in oximeter parameters | 3 months;12 months
  To assess the change in oximeter parameters: percentage of recording time with oxygen saturation < 90% (CT90), oxygen desaturation index (ODI) and mean oxygen saturation
Assessment of the degree of therapeutic adherence at 3,6 and 12 months | 3 months; 6 months;12 months
  To assess the degree of therapeutic adherence to the exercises at 3, 6 and 12 months of treatment.
Assessment of generic health-related quality of life | 3 months;12 months
  To assess the generic health-related quality of life measured by Short Form-36 Health Survey (SF-36) questionnaire
Assessment of sleep quality | 3 months;12 months
  To assess the sleep quality measured by Pittsburgh Quality of Sleep Index questionnaire
Assessment of daytime sleepiness | 3 months;12 months
  To assess the change in daytime sleepiness measured by the Epworth sleepiness scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Pneumology Department, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No